CLINICAL TRIAL: NCT04089943
Title: The Role of microRNA-210 in Regulating Oxidative Stress in Patients With Peripheral Artery Disease
Brief Title: The Role of microRNA-210 in Regulating Oxidative Stress in Patients With PAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Panagiotis Koutakis, Associate Professor, University of West Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2211301; 1R01AG064420 (NIH)
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Arterial Disease; Vascular Diseases, Peripheral; Arterial Occlusive Diseases; Atherosclerosis
Keywords: peripheral artery disease; microRNA
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Arterial Occlusive Diseases; Atherosclerosis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revascularization group (Experimental): Participants will be randomized to either an endovascular or an open bypass procedure.
  Interventions: Procedure: Revascularization operation
- Control group (Other): Healthy non-PAD participants will be recruited as control group
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Revascularization operation — Participants will be randomized into an endovascular or open bypass procedure.
  Arms: Revascularization group
Other: Control group — Healthy non-PAD participants will be recruited for the study.
  Arms: Control group

SUMMARY:
MicroRNA-210 (miR-210) can be a potential therapeutic target of patients with peripheral artery disease (PAD). Recent evidence suggests the role of miR-210 and oxidative stress in the pathophysiology of PAD and its association with mitochondrial function, oxidative metabolism, walking distances and quality of life. The protocol evaluates the mechanisms which miR-210 regulates oxidative stress and provides evidence of potential therapeutic strategies.

DETAILED DESCRIPTION:
The investigators will randomize 180 PAD patients that undergoing a revascularization operation in two groups: (1) an endovascular procedure or (2) an open bypass procedure. They are also planning to recruit 50 non-PAD healthy control subjects.

The goal is to answer the main hypothesis that miR-210 gene expression is a master regulator of oxidative stress and is associated with mitochondrial dysfunction, oxidative metabolism, walking function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. male or female 30 years or older,
2. Infrainguinal PAD,
3. critical limb ischemia, defined as arterial insufficiency with gangrene, nonhealing ischemic ulcer, or rest pain consistent,
4. candidate for both endovascular and open infra-inguinal revascularization as judged by the vascular surgeons,
5. absence of musculoskeletal (most commonly arthritis related) or neurologic (most commonly back pain and sciatica related) symptoms,
6. willingness to comply with protocol, attend follow-up appointments, complete all study assessments, and provide written informed consent.

Exclusion Criteria:

1. life expectancy of less than 2 years due to reasons other than PAD,
2. acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma,
3. current chemotherapy or radiation therapy

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
miR-210 gene expression | Change from baseline to six-month follow-up
  Measure miR-210 gene expression at baseline and after intervention
Calf muscle biopsy biochemical measures | Change from baseline to six-month follow-up
  A skeletal muscle sample will be obtained from the gastrocnemius muscle.

SECONDARY OUTCOMES:
Six-minute walk performance | Change from baseline to six-month follow-up
  Participants walking up and down a 100 foot hallway for six minutes following a standardized protocol. The goal is for them to walk as far as possible in six minutes
Graded treadmill walk performance | Change from baseline to six-month follow-up
  Participants walking on treadmill following a standardized protocol. The goal is for them to walk as far as possible while the treadmill incline increases every 2 minutes.
The 36-Item Short Form questionnaire (SF-36) | Change from baseline to six-month follow-up
  This well validated quality of life measure will be used to assess changes in patient perceived quality of life. The SF-36 is scored from 0-100, with 100 being the best score.
The Walking Impairment Questionnaire | Change from baseline to six-month follow-up
  The well validated Walking Impairment Questionnaire (WIQ) will be used to measure patient- perceived walking performance. The WIQ is scored from 0-100, with 100 being the best score.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Koutakis, PhD, Principal Investigator — University of West Florida
Locations (2):
- United States (2):
  - UT Austing Dell Medical School, Austin, Texas
  - Baylor Scott and White, Temple, Texas

IPD SHARING:
Plan to Share IPD: No